CLINICAL TRIAL: NCT02276118
Title: Comparisons of Prosthesis Fitness, Early Recovery Patterns, Functional Outcomes and Patient Satisfaction Between E.Motion-Pro, a New Mobile Bearing System and Genesis II, an Established Successful System
Brief Title: Outcome Comparison of Two Total Knee Arthroplasty Systems: e.Motion-Pro Versus Genesis II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1406/254-001
Record Dates: First submitted 2014-10-19; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- e.motion PS Pro group (Experimental): the patients who receives total knee arthroplasty with the e.motion PS pro prosthesis
  Interventions: Device: device: e.motion PS Pro
- Genesis II group (Active Comparator): the patients who receives total knee arthroplasty with the Genesis II prosthesis
  Interventions: Device: device : Genesis II

INTERVENTIONS:
Device: device: e.motion PS Pro — patients will undergo total knee arthroplasty with e.motion PS Pro implant
  Arms: e.motion PS Pro group
Device: device : Genesis II — patients will undergo total knee arthroplasty with Genesis II implant
  Arms: Genesis II group

SUMMARY:
Recently, E.Motion-PS-Pro (B.Braun-Aesculap, Tuttlingen, Germany), a new mobile bearing knee system with a unique ball and socket post-cam mechanism was developed for use in total knee arthroplasty. This study aims to determine (1) whether the use of E.Motion-PS-Pro improves prosthesis fitness for the femur and tibia in terms of under- or over-hang incidence compared to an established successful prosthesis, Genesis II (Smith & Nephew, Memphis, U.S.A.), (2) whether patients with this new prosthesis experience less pain and faster wound healing in early recovery phase, (3) whether patients with E.Motion-Pro reach functional plateaus faster than patients with Genesis II and the functional plateaus of patients with E.Motion-Pro are higher than those of patients with Genesis II.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a satisfactory treatment option for patients with advanced knee diseases that are intractable with other modalities in terms of pain relief, functional restoration, and deformity correction. Unfortunately, however, many patients have to go through a recovery period of several months during which they experience considerable pain and suffer from incompletely restored functions. In recent years, to improve the quality of life during early recovery period after TKA, great efforts have been made in multiple areas including the use of minimally invasive surgical technique, improved pain management protocols, and postoperative rehabilitation protocols. Nonetheless, this almost inevitable presence of painful and disabling recovery period is a major concern to patients scheduled for or considering TKA as a treatment option. Furthermore, this issue can become a more serious obstacle to very elderly patients who have to balance the benefits of remaining years with improved functions from replaced knees and the burden of recovery duration after TKA.

In theory, the use of a better fitting prosthesis with sound kinematic performance can shorten the duration of recovery period and improve the quality of life by reducing pain and facilitating functional recovery. Better fitting prostheses allegedly less involve prosthesis overhang at femoral condylar level, which can cause impingement symptoms and at anterior flange area, which can cause patellofemoral symptoms. Prosthesis providing better kinematic performance such as natural motion and joint stability throughout motion arc can reduce pain and discomfort in early recovery period and shorten the duration of recovery period.

Recently, E.Motion-PS-Pro (B.Braun-Aesculap, Tuttlingen, Germany), a new mobile bearing knee system with a unique ball and socket post-cam mechanism was developed. This new prosthesis was designed to achieve better prosthesis fitting, to minimize bone loss from box preparations for post-cam mechanism, to improve joint stability throughout motion arc, particularly in high flexion, and to reduce the risk for wear and fracture at the post by increasing contact area. If the intended design rationales work out well, this prosthesis shall reduce soft tissue impingement and provide better kinematic performances, which reduces pain and facilitates functional restoration.

Therefore, the current investigators aim to determine (1) whether the use of E.Motion-PS-Pro improves prosthesis fitness for the femur and tibia in terms of under- or over-hang incidence compared to an established successful prosthesis, Genesis II (Smith & Nephew, Memphis, U.S.A.), (2) whether patients with this new prosthesis experience less pain and faster wound healing in early recovery phase, (3) whether patients with E.Motion-Pro reach functional plateaus faster than patients with Genesis II and the functional plateaus of patients with E.Motion-Pro are higher than those of patients with Genesis II. The investigators hypothesize that (1) E.Motion-Pro reduces the incidence of prosthesis under- or over-hang, (2) patients with E.Motion-Pro experience less pain and faster wound healing in early recovery phase, and (3) patients with E.Motion-Pro reach functional plateau faster and the functional outcomes at 1 year are better in patients with E.Motion-Pro than those with Genesis II.

ELIGIBILITY:
Inclusion Criteria:

* patients who are decided to undergo total knee arthroplasty with diagnosis of primary osteoarthritis

Exclusion Criteria:

* the diagnosis other than primary osteoarthritis
* previous history of infection or trauma requiring surgical treatment on the knee which will receive total knee arthroplasty
* patients of 80 years or older
* patients with systemic diseases that can affect functional outcomes of TKA

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
prosthesis fit | from the start to end of surgery (expected average of 90 minutes)
  Component fitness will be evaluated by whether there is overhang (too wide or big) or underhang (too narrow or small) more than 2 mm at any of three sites: condyle, junction, and anterior flange
pain level during gait at 3 months after surgery | at 3 months after surgery
  Pain levels will be evaluated by asking how much pain patients feel during weight bearing gait at 3 months in 0-10 visual analog scale (0-no pain and 10-maximum pain)
knee swelling (circumference measured at the knee) at 3 months | at 3 months after surgery
  Knee swelling will be evaluated by measuring the leg circumference at the knee level (mid-patella), and the measured circumference will be compared with the preoperative circumference
flexion contracture and maximum flexion at 3 months | at 3 months after surgery
  Flexion contracture and further flexion will be measured by a single investigator using a 38-cm clinical goniometer with patients supine
the new American Knee Society (AKS) score at 6 months | at 6 months after surgery
  Patients will be evaluated at 6 months using the new scoring system of American Knee Society. The American Knee Society scoring system evaluates multiple aspects of outcomes: 1) Objective knee indicators (maximum points 80) - alignment (25), mediolateral (ML) stability (15), anteroposterior (AP) stability (10), range of motion (ROM) (30); 2) Knee score (maximum points 80) - symptoms (25), patient satisfaction (40), and expectation (15); 3) Function score (maximum points 100) - walking & standing (30), standard activities (30), advanced activities (25), discretionary knee activities (15)

SECONDARY OUTCOMES:
whether balanced gaps were achieved | from the start to end of surgery (expected average of 90 minutes)
  Balanced gap achievement will be called when flexion-extension and medio-lateral gaps are not beyond 2 mm difference
tourniquet time | from the start to end of surgery (expected average of 90 minutes)
  Tourniquet time will be measured as the duration in minutes from the point making skin incision to deflating tourniquet to check whether arterial bleeders are after implant fixation
blood volume drained via a vacuum drainage in the subcutaneous tissue | from the end of surgery to removal of vacuum drainage (usually at 2 days after surgery)
  blood volume drained via a vacuum drainage will be measured as the total amount drained from the end of surgery to removal of vacuum drainage in mL.
hemoglobin drop on postoperative 2 and 5 days | at 2 and 5 days after surgery
  hemoglobin drop on the 2nd and 5th postoperative days will be evaluated by subtracting hemoglobin level on the 2nd or 5th day from the preoperative level.
pain level during motion arc exercise at 2 and 6 weeks | at 2 and 6 weeks after surgery
  Pain levels during motion arc exercise will be evaluated at 2 and 6 weeks using 0-10 Visual Analogue Scale.
knee swelling at 2 and 6 weeks | at 2 and 6 weeks after surgery
  knee swelling will be evaluated at 2 and 6 weeks by noting the leg circumference at the mid-patella level
need for walking aid at 6 weeks | at 6 weeks after surgery
  Whether patients still need a walking aid (yes/no) will be noted at 6 weeks
patient satisfaction with early recovery pattern at 3 months | at 3months after surgery
  Patient satisfaction with early recovery pattern will be evaluated at 3 month using a 0-4 Likert scales (0-disappointed, 1-less satisfactory than expected, 2 - as expected, 3- more satisfactory than expected, 4 - extremely satisfactory)
flexion contracture and further flexion at 6 weeks, and 6, 12, 24 months | at 6 weeks, and 6, 12, 24 months after surgery
  Motion arc will be evaluated in extension deficit (flexion contracture) and maximum flexion at 6 weeks, 6 months, 12 months, and 2 years
patient satisfaction with replaced knees at 12 and 24 months | at 12 and 24 months after surgery
  Patients will be evaluated for their satisfaction with replaced knees at 12 and 24 months after surgery with 0-4 Likert scale and 0-10 Visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyun Kim, MD, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea